CLINICAL TRIAL: NCT01445171
Title: Surgical Treatment of Aortic Stenosis With a Next Generation Surgical Aortic Valve
Acronym: TRITON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-01
Record Dates: First submitted 2011-08-05; First posted 2011-10-03 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Aortic Valve Stenosis With Insufficiency; Aortic Valve Stenosis
Keywords: Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study Valve (Other): Subjects act as own control
  Interventions: Device: Aortic Valve Replacement with EDWARDS INTUITY Valve System

INTERVENTIONS:
Device: Aortic Valve Replacement with EDWARDS INTUITY Valve System — Aortic Valve bioprosthesis

SUMMARY:
The purpose of this clinical investigation is to confirm that the safety and performance of the EDWARDS INTUITY Valve System.

DETAILED DESCRIPTION:
This is a two-phase, non-randomized, prospective, single arm, multi-center clinical investigation. Each subject in Phase 1 and Phase 2 is consented for a period of 5 years. All subjects will be assessed for clinical follow-up at the following intervals: Discharge, 1 month, 3 months, 1 year and annually thereafter until 5 years of follow-up is achieved per subject.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* 18 years or older
* Aortic stenosis or stenosis-insufficiency of aortic valve requiring a planned replacement as indicated in the preoperative evaluation;
* Scheduled to undergo planned aortic valve replacement with or without concomitant coronary bypass surgery, MAZE procedure, septal myectomy, pacemaker/ICD implant and or atrial appendage occlusion/removal.
* Signed and dated the informed consent form prior to investigation procedures;
* Geographically stable and agrees to attend Follow up assessments at the hospital of surgical services for a maximum of 5 years.

Exclusion Criteria:

* Pure aortic insufficiency
* Requires emergency surgery
* Aneurysm of the aortic root and/or ascending aorta requiring surgical intervention
* Left ventricular ejection fraction of ≤ 25%
* Active endocarditis within 3 months prior to the scheduled aortic valve replacement surgery
* Concomitant valve (mitral, tricuspid, or pulmonic) disease requiring repair with an annuloplasty ring or replacement with prosthesis
* Prior mitral, tricuspid or pulmonic valve surgery, which included implantation of a bioprosthetic valve, mechanical valve, or annuloplasty ring.
* Myocardial infarction (MI) within 1 month prior to the scheduled aortic valve replacement surgery
* Previously implanted with EDWARDS INTUITY Aortic valve; alcohol or drug abuser
* Disease limiting life expectancy to less than 12 months
* Pregnant or lactating
* Currently participating in another drug or device clinical investigation;
* Documented blood diatheses
* Requires non-cardiac procedures such as carotid procedures or mediastinal tumor removal
* Had a stroke or transient ischemic attack (TIA) within 6-months prior to scheduled aortic valve replacement surgery
* Study site pre-operative echocardiographic assessment shows evidence of an intracardiac mass, thrombus, or vegetation
* Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days of procedure
* Documented renal insufficiency as determined by Serum creatinine ≥ 200 µmol/L (2.27 mg/dL) at screening or end-stage renal disease requiring chronic dialysis
* Documented hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2010-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Axel Haverich, Study Director — MHH Hannover
Locations (6):
- AKH Vienna-Allgemeines Krankenhaus der Stadt Wien; University Vienna, Vienna, Austria
- Germany (5):
  - Kerchoff Klinik-Bad Nauheim, Bad Nauheim
  - Herzzentrum Uniklink Koln-Klinik und Poliklinik fur Herz und Thoraxzchirurgie, Cologne
  - MHH-Medizinische Hoschschule Hannover, Hanover
  - University Leipzig: Herzzentrum Leipzig Gmbh, Leipzig
  - Klinikum der Universitat Muchen-Grosshadern; Clinic at the University of Munich, Munich

REFERENCES:
- [Result] Laufer G, Haverich A, Andreas M, Mohr FW, Walther T, Shrestha M, Rahmanian P, Holzhey D, Roth M, Schmitz C, Schramm R, Giot C, Wahlers TCW. Long-term outcomes of a rapid deployment aortic valve: data up to 5 years. Eur J Cardiothorac Surg. 2017 Aug 1;52(2):281-287. doi: 10.1093/ejcts/ezx103. PMID 28453629
- [Result] Haverich A, Wahlers TC, Borger MA, Shrestha M, Kocher AA, Walther T, Roth M, Misfeld M, Mohr FW, Kempfert J, Dohmen PM, Schmitz C, Rahmanian P, Wiedemann D, Duhay FG, Laufer G. Three-year hemodynamic performance, left ventricular mass regression, and prosthetic-patient mismatch after rapid deployment aortic valve replacement in 287 patients. J Thorac Cardiovasc Surg. 2014 Dec;148(6):2854-60. doi: 10.1016/j.jtcvs.2014.07.049. Epub 2014 Aug 1. PMID 25218544
- [Result] Kocher AA, Laufer G, Haverich A, Shrestha M, Walther T, Misfeld M, Kempfert J, Gillam L, Schmitz C, Wahlers TC, Wippermann J, Mohr FW, Roth M, Skwara A, Rahmanian P, Wiedemann D, Borger MA. One-year outcomes of the Surgical Treatment of Aortic Stenosis With a Next Generation Surgical Aortic Valve (TRITON) trial: a prospective multicenter study of rapid-deployment aortic valve replacement with the EDWARDS INTUITY Valve System. J Thorac Cardiovasc Surg. 2013 Jan;145(1):110-5; discussion 115-6. doi: 10.1016/j.jtcvs.2012.07.108. Epub 2012 Oct 8. PMID 23058665
- [Result] Wahlers TCW, Andreas M, Rahmanian P, Candolfi P, Zemanova B, Giot C, Ferrari E, Laufer G. Outcomes of a Rapid Deployment Aortic Valve Versus Its Conventional Counterpart: A Propensity-Matched Analysis. Innovations (Phila). 2018 May/Jun;13(3):177-183. doi: 10.1097/IMI.0000000000000509. PMID 29912142
- [Derived] Alaklabi AM, Abdul Rab S, Sabbah BN, Maklad AE, Dokollari A, Van den Eynde J, Pompeu Sa M, Arjomandi Rad A, Ahsan MR, Fatehi Hassanabad A. Innovations in Aortic Valve Replacement: A Comprehensive Overview of the Intuity Rapid Deployment Valve. Cardiol Rev. 2026 Jan-Feb 01;34(1):30-39. doi: 10.1097/CRD.0000000000000657. Epub 2024 Feb 9. PMID 38334371
- See also: New York Heart Association Classification — https://www.heart.org/en/health-topics/heart-failure/what-is-heart-failure/classes-of-heart-failure

RESULTS

PARTICIPANT FLOW:
Groups:
- INTUITY Aortic Valve and INTUITY Delivery System: The EDWARDS INTUITY Aortic Valve models 8300ACA and 8300ACB, and the EDWARDS INTUITY Delivery System models 8300DCA and 8300DCB are intended for use in subjects with aortic stenosis or stenosis-insufficiency requiring primary replacement of the native aortic valve.
Period: Overall Study
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Started | 295
Implanted With Study Device | 287
Completed | 200
Not Completed | 95
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 16
Not completed — Death | 51
Not completed — Subjects declined to return for followup | 9
Not completed — Consented but did not receive device | 8

BASELINE CHARACTERISTICS:
Population: The outcome is reported for subjects who received the EDWARDS INTUITY Aortic Valve models 8300ACA and 8300ACB, and the EDWARDS INTUITY Delivery System models 8300DCA and 8300DCB where data is available.
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 146
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percent of Early Adverse Events
Description: Number of early adverse events occurring within 30 days of procedure divided by the total number of enrolled subjects times 100.
Time Frame: Events occuring within 30 days of procedure
Population: The outcome is reported for subjects who received the Edwards Intuity model 8300ACA or 8300ACB device where data is available.
Measure: Number; unit: Percentage of subjects
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
Percentage of subjects
  All Cause Mortality | 1.7
  Trial Valve Related Mortality | 1.0
  Thromboembolism | 4.5
  Valve Thrombosis | 0.0
  Major Bleeding | 7.3
  All Paravalvular Leak (OPC) | 1.0
  Hemolysis | 0.7
  Endocarditis | 0.0
  Structural Valve Deterioration | 0.0
  Reoperation | 1.4
  Explant | 1.4
  Valve Related AE | 3.1

2. Primary Outcome: Percent of Late Adverse Events
Description: Number of late adverse events divided by the total number of late patient years times 100. Late patient years are calculated from 31 days post-implant to the date of the last contact (follow up or adverse event).
Time Frame: Events occurring >= 31 days and up through 5 years post-implant
Population: as for outcome 1
Measure: Number; unit: Percentage of late adverse events
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
Percentage of late adverse events
  All Cause Mortality | 3.8
  Trial Valve Related Mortality | 0.4
  Thromboembolism | 1.9
  Valve Thrombosis | 0.0
  Major Bleeding | 2.1
  All Paravalvular Leak (OPC) | 0.6
  Hemolysis | 0.2
  Endocarditis | 0.3
  Structural Valve Deterioration | 0.5
  Reoperation | 0.5
  Explant | 0.5
  Valve Related AE | 1.0

3. Other Pre Specified Outcome: Number of Subject's With Device Technical Success
Description: Device technical success is defined as the successful delivery and deployment of one bioprosthesis with one delivery system with a maximum of two attempts.
Time Frame: At time of surgery, an average of 3 hours
Population: This outcome is reported for enrolled subjects where data is available. Subjects were considered enrolled after meeting all the enrollment criteria, signing the informed consent, and after the surgeon sized the aortic annulus, and determined that the bioprosthesis could be implanted.
Measure: Count of Participants; unit: Participants
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 295
Participants | 287

4. Other Pre Specified Outcome: Number of Subject's With Procedural Success
Description: Procedure success is defined as device technical success followed by the absence of adverse events requiring device reoperation, requiring implantation of permanent pacemaker, or subject death.
Time Frame: Discharge(an average of 13 days) or 10 days post-implant, whichever comes first
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 295
Participants | 277

5. Other Pre Specified Outcome: Subject's New York Heart Association (NYHA) Functional Class Compared to Baseline
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: 1 Month, 3 Months, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 283
Participants
  1 Month: number analyzed (Participants) | 194
  1 Month: Improved | 121
  1 Month: Same | 59
  1 Month: Worsened | 14
  3 Months: number analyzed (Participants) | 262
  3 Months: Improved | 189
  3 Months: Same | 65
  3 Months: Worsened | 8
  1 Year: number analyzed (Participants) | 255
  1 Year: Improved | 191
  1 Year: Same | 57
  1 Year: Worsened | 7
  2 Years: number analyzed (Participants) | 238
  2 Years: Improved | 180
  2 Years: Same | 46
  2 Years: Worsened | 12
  3 Years: number analyzed (Participants) | 225
  3 Years: Improved | 157
  3 Years: Same | 56
  3 Years: Worsened | 12
  4 Years: number analyzed (Participants) | 207
  4 Years: Improved | 137
  4 Years: Same | 60
  4 Years: Worsened | 10
  5 Years: number analyzed (Participants) | 193
  5 Years: Improved | 125
  5 Years: Same | 52
  5 Years: Worsened | 16

6. Other Pre Specified Outcome: Subject's Average Score on the EQ-5D- Quality of Life Questionnaire Over Time
Description: The EQ-5D is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale is indexed and ranges from a minimum of 0.275 and a maximum of 1.000. A lower number indicates the participants experiences more problems and a higher number indicates the participants experiences fewer problems.
Time Frame: Baseline, 3 Months, and 1 Year post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline and 3 Months Follow-Up; Baseline and 1 Year Follow-Up: The EDWARDS INTUITY Aortic Valve models 8300ACA and 8300ACB, and the EDWARDS INTUITY Delivery System models 8300DCA and 8300DCB are intended for use in subjects with aortic stenosis or stenosis-insufficiency requiring primary replacement of the native aortic valve.
Arm/Group | Baseline and 3 Months Follow-Up | Baseline and 1 Year Follow-Up
Number analyzed (Participants) | 124 | 250
units on a scale
  Baseline | 0.79 (0.20) | 0.79 (0.19)
  Follow-Up | 0.87 (0.18) | 0.83 (0.22)

7. Other Pre Specified Outcome: Subject's Average Mean Systolic Gradient Measurements Over Time.
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: Discharge (an average of 13 days), 1 Month, 3 Months, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
mmHg
  Discharge: number analyzed (Participants) | 226
  Discharge | 10.6 (4.2)
  1 Month: number analyzed (Participants) | 10
  1 Month | 9.5 (2.8)
  3 Months: number analyzed (Participants) | 224
  3 Months | 9.0 (3.4)
  1 Year: number analyzed (Participants) | 230
  1 Year | 9.0 (3.5)
  2 Years: number analyzed (Participants) | 92
  2 Years | 8.8 (3.0)
  3 Years: number analyzed (Participants) | 186
  3 Years | 9.6 (4.3)
  4 Years: number analyzed (Participants) | 136
  4 Years | 10.0 (4.7)
  5 Years: number analyzed (Participants) | 161
  5 Years | 9.9 (5.1)

8. Other Pre Specified Outcome: Subject's Average Effective Orifice Area Measurements Over Time.
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Discharge (an average of 13 days), 1 Month, 3 Months, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Centimeters Squared
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
Centimeters Squared
  Discharge: number analyzed (Participants) | 178
  Discharge | 1.7 (0.2)
  1 Month: number analyzed (Participants) | 10
  1 Month | 1.6 (0.2)
  3 Months: number analyzed (Participants) | 204
  3 Months | 1.7 (0.2)
  1 Year: number analyzed (Participants) | 211
  1 Year | 1.7 (0.2)
  2 Years: number analyzed (Participants) | 81
  2 Years | 1.7 (0.2)
  3 Years: number analyzed (Participants) | 178
  3 Years | 1.7 (0.2)
  4 Years: number analyzed (Participants) | 134
  4 Years | 1.7 (0.3)
  5 Years: number analyzed (Participants) | 151
  5 Years | 1.7 (0.3)

9. Other Pre Specified Outcome: Subject's Amount of Aortic Valvular Regurgitation Over Time
Description: Aortic valvular regurgitation occurs when the aortic valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Aortic valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation.
Time Frame: Discharge (an average of 13 days), 1 Month, 3 Months, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
Participants
  Discharge: number analyzed (Participants) | 257
  Discharge: 0 None/+1 Trivial | 244
  Discharge: +2 Mild | 10
  Discharge: +3 Moderate | 2
  Discharge: +4 Severe | 1
  1 Month: number analyzed (Participants) | 11
  1 Month: 0 None/+1 Trivial | 10
  1 Month: +2 Mild | 1
  1 Month: +3 Moderate | 0
  1 Month: +4 Severe | 0
  3 Months: number analyzed (Participants) | 251
  3 Months: 0 None/+1 Trivial | 235
  3 Months: +2 Mild | 11
  3 Months: +3 Moderate | 4
  3 Months: +4 Severe | 1
  1 Year: number analyzed (Participants) | 248
  1 Year: 0 None/+1 Trivial | 231
  1 Year: +2 Mild | 14
  1 Year: +3 Moderate | 3
  1 Year: +4 Severe | 0
  2 Years: number analyzed (Participants) | 97
  2 Years: 0 None/+1 Trivial | 86
  2 Years: +2 Mild | 7
  2 Years: +3 Moderate | 4
  2 Years: +4 Severe | 0
  3 Years: number analyzed (Participants) | 193
  3 Years: 0 None/+1 Trivial | 177
  3 Years: +2 Mild | 12
  3 Years: +3 Moderate | 4
  3 Years: +4 Severe | 0
  4 Years: number analyzed (Participants) | 140
  4 Years: 0 None/+1 Trivial | 125
  4 Years: +2 Mild | 11
  4 Years: +3 Moderate | 4
  4 Years: +4 Severe | 0
  5 Years: number analyzed (Participants) | 174
  5 Years: 0 None/+1 Trivial | 161
  5 Years: +2 Mild | 9
  5 Years: +3 Moderate | 4
  5 Years: +4 Severe | 0

10. Other Pre Specified Outcome: Subject's Average White Blood Cell Count Measurement Over Time.
Description: Laboratory analysis of White Blood Cell Count on blood drawn from subject; WBC fight infection.
Time Frame: Baseline, 3 Months, 1 Year, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliters
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
10^3 cells/microliters
  Baseline: number analyzed (Participants) | 285
  Baseline | 6.80 (2.0)
  3 Months: number analyzed (Participants) | 257
  3 Months | 6.97 (1.8)
  1 Year: number analyzed (Participants) | 251
  1 Year | 7.10 (2.0)
  5 Years: number analyzed (Participants) | 176
  5 Years | 7.31 (2.0)

11. Other Pre Specified Outcome: Subject's Average Red Blood Cells Count Over Time.
Description: Laboratory Analysis of Red Blood Cell Count on blood drawn from subjects; RBC carry oxygen.
Time Frame: Baseline, 3 Months, 1 Year, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliters
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
10^6 cells/microliters
  Baseline: number analyzed (Participants) | 285
  Baseline | 4.30 (0.5)
  3 Months: number analyzed (Participants) | 257
  3 Months | 4.40 (0.5)
  1 Year: number analyzed (Participants) | 251
  1 Year | 4.36 (0.5)
  5 Years: number analyzed (Participants) | 176
  5 Years | 4.35 (0.8)

12. Other Pre Specified Outcome: Subject's Average Hemoglobin Count Over Time.
Description: Laboratory Analysis of Hemoglobin Count on blood drawn from subjects. Hemoglobin is an oxygen-carrying protein in red blood cells.
Time Frame: Baseline, 3 Months, 1 Year, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
g/dl
  Baseline: number analyzed (Participants) | 286
  Baseline | 12.87 (1.7)
  3 Months: number analyzed (Participants) | 257
  3 Months | 12.49 (1.4)
  1 Year: number analyzed (Participants) | 251
  1 Year | 13.00 (1.5)
  5 Years: number analyzed (Participants) | 176
  5 Years | 13.16 (1.6)

13. Other Pre Specified Outcome: Subject's Average Hematocrit Percentage Over Time.
Description: Laboratory Analysis of Hematocrit Percentage on blood drawn from subjects. Hematocrit is the proportion of red blood cells to the fluid component (plasma) in the blood.
Time Frame: Baseline, 3 Months, 1 Year, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
percentage of red blood cells
  Baseline: number analyzed (Participants) | 285
  Baseline | 38.29 (4.7)
  3 Months: number analyzed (Participants) | 257
  3 Months | 38.07 (4.1)
  1 Year: number analyzed (Participants) | 251
  1 Year | 38.93 (4.1)
  5 Years: number analyzed (Participants) | 176
  5 Years | 39.58 (4.4)

14. Other Pre Specified Outcome: Subject's Average Platelet Count Over Time.
Description: Laboratory Analysis of Platelet Count on blood drawn from subjects; platelets help with blood clotting.
Time Frame: Baseline, 3 Months, 1 Year, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^3 platelets per microliter
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
10^3 platelets per microliter
  Baseline: number analyzed (Participants) | 286
  Baseline | 220.33 (66.30)
  3 Months: number analyzed (Participants) | 256
  3 Months | 223.07 (59.70)
  1 Year: number analyzed (Participants) | 251
  1 Year | 213.22 (60.40)
  5 Years: number analyzed (Participants) | 176
  5 Years | 206.85 (63.5)

15. Other Pre Specified Outcome: Subject's Average Reticulocytes Percentage Over Time.
Description: Reticulocytes are immature red blood cells; a reticulocyte blood test measures the amount of these cells in the blood.
Time Frame: Baseline, 3 Months, 1 Year, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of reticulocytes
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
percentage of reticulocytes
  Baseline: number analyzed (Participants) | 194
  Baseline | 2.13 (2.5)
  3 Months: number analyzed (Participants) | 250
  3 Months | 1.59 (1.9)
  1 Year: number analyzed (Participants) | 249
  1 Year | 2.07 (5.0)
  5 Years: number analyzed (Participants) | 166
  5 Years | 1.82 (2.2)

16. Other Pre Specified Outcome: Subject's Average Haptoglobin Measurement Over Time.
Description: Laboratory Analysis of Haptoglobin on blood drawn from subjects; Haptoglobin is a protein produced by the liver.
Time Frame: Baseline, 3 Months, 1 Year, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
g/L
  Baseline: number analyzed (Participants) | 202
  Baseline | 63.08 (69.50)
  3 Months: number analyzed (Participants) | 249
  3 Months | 82.15 (81.10)
  1 Year: number analyzed (Participants) | 250
  1 Year | 80.65 (80.50)
  5 Years: number analyzed (Participants) | 172
  5 Years | 79.36 (81.20)

17. Other Pre Specified Outcome: Subject's Average Serum LDH Measurement Over Time.
Description: The lactate dehydrogenase (LDH) test looks for signs of damage to the body's tissues.
Time Frame: Baseline, 3 Months, 1 Year, and 5 Years post-implant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
Number analyzed (Participants) | 287
U/L
  Baseline: number analyzed (Participants) | 274
  Baseline | 223.91 (53.0)
  3 Months: number analyzed (Participants) | 242
  3 Months | 271.37 (87.20)
  1 Year: number analyzed (Participants) | 247
  1 Year | 250.56 (76.20)
  5 Years: number analyzed (Participants) | 169
  5 Years | 254.46 (76.30)

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through five years post-implant
Description: The outcome is reported for subjects who received the Edwards Intuity model 8300ACA or 8300ACB device where data is available.
Arm/Group | INTUITY Aortic Valve and INTUITY Delivery System
All-Cause Mortality (participants affected / at risk) | 51/287
Serious Adverse Events (participants affected / at risk) | 233/287
Other Adverse Events (participants affected / at risk) | 189/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTUITY Aortic Valve and INTUITY Delivery System (N=287)
Other (General disorders) | 137 (206)
Pulmonary - Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 57 (60)
Infection - Other (Infections and infestations) | 37 (45)
Cardiac - Other (Cardiac disorders) | 32 (35)
Gastrointestinal - Other (Gastrointestinal disorders) | 26 (34)
Cardiac - Atrial Fibrillation (Cardiac disorders) | 32 (32)
Other - Anemia (General disorders) | 25 (27)
Cardiac - Heart Failure (Cardiac disorders) | 20 (26)
Cardiac - Other Arrhythmia (Cardiac disorders) | 18 (18)
Cardiac - AV Block III (Cardiac disorders) | 17 (17)
Embolic Event - Stroke (Cardiac disorders) | 16 (17)
Infection - Local (Infections and infestations) | 16 (17)
Infection - Pneumonia (Infections and infestations) | 16 (17)
Renal - Renal Failure (Renal and urinary disorders) | 13 (14)
Vascular - Other (Vascular disorders) | 12 (14)
Bleeding - Gastrointestinal (Blood and lymphatic system disorders) | 10 (13)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Bleeding - Post-Procedural (Blood and lymphatic system disorders) | 12 (12)
Bleeding - Other (Blood and lymphatic system disorders) | 11 (12)
Cardiac - Hypertension (Cardiac disorders) | 11 (11)
Pulmonary - Respiratory Dysfunction/Insufficiency (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Renal - Renal Dysfunction (Renal and urinary disorders) | 9 (9)
Cardiac - Atrial Flutter (Cardiac disorders) | 8 (8)
Cardiac - Pericardial Effusion (Cardiac disorders) | 8 (8)
Embolic Event - TIA (Cardiac disorders) | 7 (7)
Infection - Sternal Wound Infection (Infections and infestations) | 5 (7)
Cardiac - Cardiac Arrest (Cardiac disorders) | 6 (6)
Cardiac - Myocardial Infarction (Cardiac disorders) | 6 (6)
Infection - Sepsis/Septicemia (Infections and infestations) | 6 (6)
Cardiac - Angina, Stable (Cardiac disorders) | 5 (6)
Pulmonary - Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Infection - Bacteremia (Infections and infestations) | 5 (5)
Pulmonary - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Renal - Other (Renal and urinary disorders) | 5 (5)
Cardiac - Angina, Unstable (Cardiac disorders) | 4 (5)
Bleeding - Anticoagulant Related (Blood and lymphatic system disorders) | 4 (4)
Bleeding - Hematoma (Blood and lymphatic system disorders) | 4 (4)
Bleeding - Pericardial Tamponade (Blood and lymphatic system disorders) | 4 (4)
Cardiac - Bradycardia (Cardiac disorders) | 4 (4)
Other - Allergic Reaction (General disorders) | 4 (4)
Vascular - Deep Vein Thrombosis (DVT) (Cardiac disorders) | 4 (4)
Infection - Endocarditis (Aortic Valve) (Infections and infestations) | 3 (3)
Bleeding - Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Bleeding - Procedural (Blood and lymphatic system disorders) | 2 (2)
Cardiac - Hypotension (Cardiac disorders) | 2 (2)
Cardiac - Supraventricular Tachycardia (SVT) (Cardiac disorders) | 2 (2)
Embolic Event - Other (Blood and lymphatic system disorders) | 2 (2)
Embolic Event - Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hepatic - Other (Hepatobiliary disorders) | 2 (2)
Multisystem Organ Failure (General disorders) | 2 (2)
Valvular - Paravalvular Leak - Moderate (Cardiac disorders) | 2 (2)
Bleeding - Intracranial (Blood and lymphatic system disorders) | 1 (1)
Cardiac - Aortic Dissection - Type A (Cardiac disorders) | 1 (1)
Cardiac - Aortic Dissection - Type B (Cardiac disorders) | 1 (1)
Cardiac - AV Block II (Cardiac disorders) | 1 (1)
Cardiac - Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cardiac - Pericardial Tamponade (Cardiac disorders) | 1 (1)
Cardiac - Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Embolic Event - Peripheral Embolic Event (Cardiac disorders) | 1 (1)
Hepatic - Liver Failure (Hepatobiliary disorders) | 1 (1)
Infection - Endocarditis (Mitral Valve) (Infections and infestations) | 1 (1)
Infection - Systemic (Infections and infestations) | 1 (1)
Pulmonary - Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary - Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary - Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Valvular - Aortic Regurgitation - Moderate-Severe (Cardiac disorders) | 1 (1)
Valvular - Mitral Regurgitation - Mild-Moderate (Cardiac disorders) | 1 (1)
Valvular - Mitral Regurgitation - Moderate-Severe (Cardiac disorders) | 1 (1)
Valvular - Other Mitral Valve (Cardiac disorders) | 1 (1)
Valvular - Paravalvular Leak - Mild (Cardiac disorders) | 1 (1)
Vascular - Vascular Access Site Complication (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTUITY Aortic Valve and INTUITY Delivery System (N=287)
Other (General disorders) | 85 (128)
Infection - Other (Infections and infestations) | 45 (50)
Cardiac - Atrial Fibrillation (Cardiac disorders) | 43 (43)
Gastrointestinal - Other (Gastrointestinal disorders) | 12 (17)
Pulmonary - Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Infection - Local (Infections and infestations) | 13 (14)
Other - Anemia (General disorders) | 11 (11)
Cardiac - BBB - Left Complete (Cardiac disorders) | 9 (9)
Renal - Renal Dysfunction (Renal and urinary disorders) | 9 (9)
Valvular - Mitral Regurgitation - Mild (Cardiac disorders) | 9 (9)
Cardiac - Other (Cardiac disorders) | 8 (8)
Cardiac - BBB - Left Partial (Cardiac disorders) | 7 (7)
Cardiac - Other Arrhythmia (Cardiac disorders) | 7 (7)
Infection - Pneumonia (Infections and infestations) | 7 (7)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Cardiac - Atrial Flutter (Cardiac disorders) | 6 (6)
Infection - Sternal Wound Infection (Infections and infestations) | 6 (6)
Renal - Other (Renal and urinary disorders) | 5 (5)
Valvular - Aortic Regurgitation - Mild (Cardiac disorders) | 5 (5)
Bleeding - Hematoma (Blood and lymphatic system disorders) | 4 (4)
Bleeding - Other (Blood and lymphatic system disorders) | 4 (4)
Cardiac - BBB - Right Complete (Cardiac disorders) | 4 (4)
Infection - Bacteremia (Infections and infestations) | 4 (4)
Vascular - Deep Vein Thrombosis (DVT) (Cardiac disorders) | 4 (4)
Other - Allergic Reaction (General disorders) | 3 (4)
Bleeding - Anticoagulant Related (Blood and lymphatic system disorders) | 3 (3)
Cardiac - AV Block I (Cardiac disorders) | 3 (3)
Cardiac - Bradycardia (Cardiac disorders) | 3 (3)
Cardiac - Hypertension (Cardiac disorders) | 3 (3)
Cardiac - Ventricular Tachycardia (Cardiac disorders) | 3 (3)
Hepatic - Other (Gastrointestinal disorders) | 3 (3)
Valvular - Aortic Stenosis - Moderate (Cardiac disorders) | 3 (3)
Bleeding - Gastrointestinal (Blood and lymphatic system disorders) | 2 (2)
Cardiac - AV Block III (Cardiac disorders) | 2 (2)
Cardiac - Pericardial Effusion (Cardiac disorders) | 2 (2)
Embolic Event - Other (Blood and lymphatic system disorders) | 2 (2)
Embolic Event - Stroke (Blood and lymphatic system disorders) | 2 (2)
Embolic Event - TIA (Blood and lymphatic system disorders) | 2 (2)
Bleeding - Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Heparin Induced Thrombocytopenia (HITS) (Blood and lymphatic system disorders) | 1 (1)
Cardiac - Angina, Stable (Cardiac disorders) | 1 (1)
Cardiac - Heart Failure (Cardiac disorders) | 1 (1)
Cardiac - Hypotension (Cardiac disorders) | 1 (1)
Cardiac - Supraventricular Tachycardia (SVT) (Cardiac disorders) | 1 (1)
Embolic Event - Peripheral Embolic Event (Blood and lymphatic system disorders) | 1 (1)
Infection - Systemic (Infections and infestations) | 1 (1)
Pulmonary - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary - Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary - Respiratory Dysfunction/Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary - Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Valvular - Aortic Regurgitation - Mild-Moderate (Cardiac disorders) | 1 (1)
Valvular - Aortic Stenosis - Mild (Cardiac disorders) | 1 (1)
Valvular - Aortic Stenosis - Severe (Cardiac disorders) | 1 (1)
Valvular - Mitral Regurgitation - Moderate-Severe (Cardiac disorders) | 1 (1)
Valvular - Other Mitral Valve (Cardiac disorders) | 1 (1)
Valvular - Other Tricuspid Valve (Cardiac disorders) | 1 (1)
Valvular - Paravalvular Leak - Mild/Moderate (Cardiac disorders) | 1 (1)
Valvular - Paravalvular Leak - Moderate (Cardiac disorders) | 1 (1)
Valvular - Paravalvular Leak - Trace/Trivial (Cardiac disorders) | 1 (1)
Valvular - Structural Deterioration (Cardiac disorders) | 1 (1)
Valvular - Tricuspid Regurgitation (Cardiac disorders) | 1 (1)
Vascular - Other (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of overall study results which have not been released requires written approval of Sponsor, but presentation of site-specific results can occur subject to review by Sponsor. Manuscripts will be submitted to Sponsor for review 60 days prior to submission of manuscript for publication/presentation. Sponsor may ask for a 90 day delay of submission of manuscripts for publication to protect proprietary information and filing of related patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-09-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT01445171/Prot_SAP_000.pdf